CLINICAL TRIAL: NCT05574335
Title: A T Cell Phenotype Signature Driven Dose Finding Study With Siplizumab in Type 1 Diabetes Mellitus (ITN095AI)
Brief Title: Siplizumab in T1DM
Acronym: DESIGNATE
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Prior to termination the DESIGNATE study was an on enrollment hold due to greater than anticipated lymphodepletion. The pharmaceutical partner decided not to reopen its own T1D trial and ceased development of siplizumab in autoimmunity.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAIT ITN095AI
Record Dates: First submitted 2022-09-19; First posted 2022-10-10 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: diabetic; Type 1 diabetes; T1DM; siplizumab
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — siplizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Adults with T1D 0.08 mg/kg SQ dose (Experimental): Cohort 1 Group1: 0.08 mg/kg SQ dose for a total of 12 weeks
  Interventions: Drug: Siplizumab
- Adults with T1D 0.12 mg/kg SQ dose (Experimental): Cohort 1 Group 2: 0.12 mg/kg SQ dose for a total of 12 weeks
  Interventions: Drug: Siplizumab
- Adults with T1D 0.18 mg/kg SQ dose (Experimental): Cohort 1 Group 3:0.18 mg/kg SQ dose for a total of 12 weeks
  Interventions: Drug: Siplizumab
- Adults with T1D 0.22 mg/kg SQ dose (Experimental): Cohort 1 Group 4: 0.22 mg/kg SQ dose for a total of 12 weeks
  Interventions: Drug: Siplizumab
- Children with T1D 0.08 mg/kg SQ dose (Experimental): Cohort 2 Group 1:0.08 mg/kg SQ dose for a total of 12 weeks
  Interventions: Drug: Siplizumab
- Children with T1D 0.12 mg/kg SQ dose (Experimental): Cohort 2 Group 2:0.12 mg/kg SQ dose for a total of 12 weeks
  Interventions: Drug: Siplizumab
- Children with T1D 0.18 mg/kg SQ dose (Experimental): Cohort 2 Group 3: 0.18 mg/kg SQ dose for a total of 12 weeks
  Interventions: Drug: Siplizumab
- Children with T1D 0.22 mg/kg SQ dose (Experimental): Cohort 2 Group 4: 0.22 mg/kg SQ dose for a total of 12 weeks
  Interventions: Drug: Siplizumab

INTERVENTIONS:
Drug: Siplizumab — Weekly siplizumab doses for a total of 12 weeks
  Other Names: TCD 601

SUMMARY:
This is a multicenter, Phase Ib, open-label, siplizumab dose-finding study in individuals aged 8-45 years with a Type 1 diabetes mellitus (T1DM) diagnosis. within 18 months of V0. Participants will be randomized 1:1:1:1 to one of four possible siplizumab dosing arms. All dosing arms will receive weekly siplizumab doses for a total of 12 weeks. After the completion of treatment, participants will undergo follow-up visits at weeks 12, 24, 36 and 52 which include longitudinal MMTTs. If indicated, participants will enter into long-term safety monitoring for up to an additional 48 weeks. Blood samples for mechanistic analyses will be obtained during the treatment phase and thereafter. Adults aged 18- 45 will be enrolled initially at the study sites.

The primary objective is to identify a safe, metabolically favorable, dosing regimen for siplizumab in patients with type 1 diabetes that induces changes in T cell phenotypes observed with alefacept therapy in new-onset T1DM.

The secondary objectives are to:

1. Assess the safety profile of siplizumab in recently diagnosed T1DM.
2. Assess the effects of siplizumab on residual beta cell function in recently diagnosed T1DM participants.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide informed consent (parental permission and informed assent of minor, if applicable).
2. Male or female between 8 to 45 years of age.
3. Diagnosis of T1DM within 18 months (550 days) of enrollment (V0).
4. Positive for at least one diabetes-related autoantibody, including:

   1. Glutamate decarboxylase (GAD-65),
   2. Insulin, if obtained within 10 days of the onset of exogenous insulin therapy,
   3. Insulinoma antigen-2 (IA-2), or
   4. Zinc transporter-8 (ZnT8).
5. Peak stimulated C-peptide level > 0.15 nmol/L following a MMTT conducted ≥ 21 days from diagnosis and within 37 days of enrollment (V0).
6. Completion of a SARS-CoV-2 vaccination, according to current CDC recommendations and FDA approval(s) or emergency use authorization(s). If the participant requires administration of vaccine(s) to meet eligibility requirements, they must complete the vaccination series at least 2 weeks prior to enrollment (V0).

Exclusion Criteria:

1. 1. Use of investigational drugs within 24 weeks of participation with the exception of any vaccine for the prevention of SARS-CoV-2 infection and emergency use authorization medications for treating SARS-CoV-2.
2. Severe reaction or anaphylaxis to humanized monoclonal antibodies.
3. Inability to complete a mixed meal tolerance test:

   1. History of significant allergy (e.g., anaphylaxis) to milk or soy proteins.
   2. Inability to disable hybrid closed loop system.
4. History of recent (within 180 days of V0) or ongoing uncontrolled bacterial, viral, fungal or other opportunistic infections, including:

   1. Human immunodeficiency virus (HIV),
   2. Current or prior infection with hepatitis B (HBV), as indicated by positive HBsAg or positive HBcAb,
   3. Current or prior hepatitis C (HCV), unless treated with anti-viral therapy with achievement of a sustained virologic response (undetectable viral load 12 weeks after cessation of therapy),
   4. Positive QuantiFERON-TB Gold or QuantiFERON-TB Gold Plus tests. PPD or T-SPOT®.TB may be substituted for the QuantiFERON-TB Gold or QuantiFERON-TB Gold Plus tests,
   5. Active infection with EBV as detected by PCR or serology at the screening visit (V-1),
   6. Active infection with cytomegalovirus (CMV) as detected by PCR or serology at the screening visit (V-1),
5. Positive molecular testing of SARS-CoV-2 within 30 days of V-1.
6. Any of the following laboratory abnormalities confirmed by repeat tests at least 1 week apart:

   1. White blood count (WBC) < 3 x 103/μL;,
   2. CD 3+ CD4+, T cell count below the lower limit of normal,
   3. Platelet count < 150,000 /μL,
   4. Hemoglobin < 10 g/dL,
   5. ALT ≥ 2x upper limit of normal (ULN) or
   6. AST ≥ 2x ULN
   7. Serum creatinine >1.5x ULN in adults or >ULN in pediatrics.
   8. Absolute lymphocyte count (ALC) below the LLN.
7. Prior or current treatment that is known to alter the natural history of T1DM or immunologic status, including high dose inhaled, extensive topical or systemic glucocorticoids.
8. Current or prior (within last 14 days of the V-1 MMTT) use of any medication known to influence glucose tolerance (e.g., atypical antipsychotics, diphenylhydantoin, thiazide, or other potassium-depleting diuretics, β-adrenergic blockers, niacin).
9. Current or prior (within the last 30 days of the V-1 MMTT) use of non-insulin medications to treat insulin resistance or elevated glucose levels.
10. Previous or current diagnosis of malignancy.
11. History of bone marrow transplantation, solid organ transplantation, or primary immunodeficiencies.
12. History or diagnoses of other autoimmune diseases with the exception of stable thyroid or celiac disease.
13. History of significant cardiovascular disease.
14. Vaccination with a live attenuated vaccine (e.g., varicella, measles, mumps, rubella, cold-attenuated intranasal influenza vaccine, bacillus Calmette- Guérin, and smallpox) within 30 days of V0.
15. Women of child-bearing potential who are unwilling to use a medically acceptable form of contraception from 14 days prior to V0 until study Week 52.
16. Women who are pregnant, lactating, or planning on pregnancy during the study.
17. Current, diagnosed mental illness (e.g., severe depression), current diagnosed or self-reported drug, or alcohol abuse that, in the opinion of the investigator, would interfere with the participant's ability to comply with study requirements.
18. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.

Ages: 8 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2023-04-26 (Actual); Primary Completion 2025-05-14 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
Number of Participants with a T cell phenotype signature response | From week 0 (baseline) to week 12
  Evaluating four siplizumab dosing regimens for induction of a T cell phenotype signature is based on a 20% increase or greater from baseline in PD1+TIGIT+ frequency within circulating CD4 Tem and a 75% increase or greater from baseline in the CD4 Treg/Tem ratio in blood.
  The two criteria will be evaluated at weeks 2, 4, 8, and 12. An individual who achieves both signature criteria at any time point on or before week 12 is counted as having the signature response. Both criteria do not need to be achieved at the same time point.

SECONDARY OUTCOMES:
Frequency of Adverse Events (AEs) in all siplizumab dosing arms | From week 0 to week 52
  AE will include any untoward medical occurrence associated with siplizumab administration or any study-mandated procedure
Mixed Meal Tolerance Test (MMTT)-stimulated mean 2-hour C-peptide AUC | At Week 12, 24, 36, 52
  The mean 2-hour C-peptide AUC, measured in nmol/L, is computed by dividing the total AUC by 120 minutes
Insulin use (U/kg/day) | At Weeks 12, 24, 36 and 52.
  Measured as U/kg body weight/day; participants should record the type and amount of insulin they have used during the 5-day period immediately preceding the beginning of treatment, middle of treatment, end of treatment, and at all follow-up visits

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Gitelman, M.D., Study Chair — University of California San Francisco, School of Medicine: Diabetes Center
Locations (5):
- United States (5):
  - University of Colorado School of Medicine: Barbara Davis Center for Diabetes, Aurora, Colorado
  - University of Iowa Children's Hospital: Department of Pediatrics, Pediatric Endocrinology and Diabetes, Iowa City, Iowa
  - Columbia University Medical Center: Naomi Berrie Diabetes Center, New York, New York
  - University of Texas Southwestern Medical Center: Department of Internal Medicine, Division of Endocrinology, Dallas, Texas
  - Benaroya Research Institute at Virginia Mason: Diabetes Research Program, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.
Time Frame: On average, within 24 months after database lock for the trial.
Access Criteria: Open access.
URL: https://www.immport.org/home

REFERENCES:
- See also: Immune Tolerance Network (ITN) — https://www.immunetolerance.org/
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait